CLINICAL TRIAL: NCT06620601
Title: Diagnosis and Treatment of Sleep Apnea in Shelter Residents
Brief Title: Digital Technology for Sleep and Homelessness
Acronym: HNSLEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Azadeh Yadollahi, Senior Scientist and Associate Professor, University Health Network, Toronto
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-5862
Record Dates: First submitted 2024-08-06; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sleep Apnea; Sleep Disorder; Sleep Deprivation; Sleep Disturbance
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Wake Disorders; Sleep Deprivation; Parasomnias | interventions — Therapeutics; Occlusal Splints; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diagnosis (Experimental): Description:
  A portable polysomnography device to assess sleep apnea in individuals at risk of sleep apnea. The Prodigy 2 has Health Canada Approval for home sleep study. The system is small, easy to use, and can be setup by a research technician at the shelter. Prodigy measures thoraco-abdominal motion, nasal airflow, oxyhemoglobin saturation (SpO2), cardiac function with electrocardiogram and leg movement. The main advantage of Prodigy 2 to other portable devices is that it has a simple headband to record forehead electroencephalogram to detect rapid eye movement (REM) and non-REM sleep stages. After processing Prodigy 2 signals, an apnea-hypopnea index (AHI) will be calculated for each participant based on the number of respiratory events (apneas or hypopneas) per hour of sleep. The investigators will measure AHI, REM AHI, non-REM AHI, AHI in different body postures, snoring duration, arousal index, sleep time with SpO2<90%, oxygen desaturation index (ODI), and sleep efficiency.
  Interventions: Diagnostic Test: Portable Polysomnography; Other: Questionnaires
- Treatment (Experimental): Description:
  Individuals who are diagnosed with sleep apnea, and are deemed eligible for treatment, will receive a treatment option based on Canadian Agency for Drugs and Technologies in Health (CADTH), physician recommendations, and the participant's preferences. In this study, auto-titrating positive airway pressure (Auto-CPAP) and Mandibular advancement device (MAD) will be the main modalities of treatment.
  Interventions: Device: Treatment; Other: Questionnaires
- Screening (Other): Also, the participants are asked to complete the following questionnaires with the help of a research assistant. The result of the application will be combined with the questionnaires for the final risk assessment.
  * Participant Demographics questionnaire
  * STOP-Bang
  * Insomnia severity index
  * Epworth sleepiness score (ESS)
  * Functional outcome of Sleep Questionnaire (FOSQ-10)
  * Beck Depression Inventory (BDI)
  * Chalder Fatigue Scale (CFQ)
  * Health Information Technology Usability Evaluation Scale (Health-ITUES) Questionnaire
  * Oral Health Impact Profile - 14 (OHIP-14)
  * Asthma Control Test (ACT)
  * Primary care post-traumatic stress disorder (PTSD) screen (PC-PTSD-5)
  * A survey to help identify barriers to treatment in the people experiencing homelessness (General Survey)
  Interventions: Other: Questionnaires

INTERVENTIONS:
Diagnostic Test: Portable Polysomnography — Research assistants set up the portable polysomnography (Prodigy) for the overnight sleep study.
  Arms: Diagnosis
Device: Treatment — Based on the decision aid, patient preference, and CADTH recommendations, the sleep physicians will recommend the participant to use Auto-CPAP or MAD for six months.
  Other Names: Continous Positive Airway Pressure; Mandibular advancement device
  Arms: Treatment
Other: Questionnaires — Participants will complete eleven questionnaires: Stop-Bang, Insomnia severity index, Epworth sleepiness score (ESS), quality of life (FOSQ-10), Beck Depression Inventory (BDI), Chalder Fatigue Scale (CFQ), primary care post-traumatic stress disorder (PTSD) scale (PC-PTSD-5), Asthma control questionnaire (ACQ), OHIP-14, and Participant demographics. The RA will help the participants complete the questionnaires (~one and a half hours in total).

SUMMARY:
In Canada, 35,000 people are experiencing homelessness on any night. Compared to the general population, people experiencing homelessness (PEH) sleep less and experience increased daytime fatigue. A common sleep disorder and treatable cause of morbidity and low quality of life is sleep apnea. High prevalence of chronic comorbid disorders of sleep apnea in PEH suggest high prevalence of sleep apnea, but the rate of sleep apnea treatment in PEH is very low. Also, in PEH, individual and systemic barriers lead to a high rate of underdiagnosed and untreated sleep apnea. Mortality is higher in PEH than the general population, and sleep apnea remains a potential silent cause of morbidity and low quality of life in PEH. Our goal is to diagnose and treat sleep apnea in people living in shelters and to examine the effect of patient-centered treatment on their quality of life.

DETAILED DESCRIPTION:
Background:

Disadvantaged individuals, including people experiencing homelessness, are at higher risk of getting infected, transmitting disease, and having poor health outcomes. Access to medical care, even within a system of universal health insurance like that of Canada, is decreased among people experiencing homelessness, but available evidence has demonstrated the efficacy of using telemedicine to reach vulnerable people in remote areas or people experiencing homelessness. However, at present, telemedicine-facilitated care in Canada is predominantly devoid of any technology to evaluate patient vital signals. The application of such technology to this population, if feasible, could have transformational implications for monitoring and management of such disadvantaged populations. Currently, it is known that there is a greater prevalence of chronic health diseases such as asthma, cardiology, and respiratory diseases in people experiencing homelessness. But there is no literature on the prevalence of obstructive sleep apnea (OSA) in the people experiencing homelessness. OSA is a condition characterized by repeated episodes of breathing cessation during sleep. Patients with OSA can suffer from daytime sleepiness, fatigue, and lack of energy. OSA is also associated with the conditions that account for the leading causes of mortality in adults: hypertension, cardiovascular, and cerebrovascular diseases. Seeing as the people experiencing homelessness already face many societal barriers to healthcare access, it is likely that there may exist a higher prevalence of undiagnosed OSA among the people experiencing homelessness.

Rationale:

From past studies, chronic diseases have been shown to be of higher prevalence in the people experiencing homelessness versus the general population, with an emphasis on a high prevalence of asthma and hypertension in the people experiencing homelessness. There is already a well-established connection between the prevalence of OSA in patients who have asthma and/or hypertension and OSA is already a highly undiagnosed condition in the general population. OSA also contributes to many other chronic health conditions. Given the strong association of hypertension and asthma with OSA, and the above average prevalence of both asthma and hypertension, among other chronic diseases, in this population, it is reasonable to infer that there might also be a high prevalence of undiagnosed OSA among the people experiencing homelessness. The use of technology and telemedicine will decrease the barriers in receiving care for people experiencing homelessness and allow for ease of access to diagnose OSA.

Inclusion/Exclusion Criteria:

The eligibility criteria for participants will include residing in a shelter at the time of recruitment, and being >18 years old. Participants with allergies to medical tape will be excluded from the study. For treatment protocol, exclusion criteria for mandibular advancement treatment will be dental and oral health requiring extensive dental treatment or periodontal disease with tooth mobility.

Hypotheses:

The investigators hypothesize that the prevalence of obstructive sleep apnea in the people experiencing homelessness will exceed that observed in the general population, as do the associated conditions of hypertension and asthma. Furthermore, the investigators hypothesize that the use of technology will help to decrease barriers in diagnosing and providing treatment for OSA.

Primary Objectives:

1. Assess the prevalence of sleep apnea in shelter residents
2. Evaluate the effects of preferred sleep apnea treatment on quality of life of the people experiencing homelessness

Significance:

The investigators anticipate the results of this study to help lower barriers to healthcare and provide better health outcomes for people experiencing homelessness. This study will provide insight into the prevalence of OSA in people experiencing homelessness and the feasibility of using technology in telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Residing in a shelter at the time of recruitment
* Age >18 years old

Exclusion Criteria:

* Allergies to medical tape [for diagnosis study].
* Requiring extensive dental treatment or periodontal disease with tooth mobility [for treatment study].

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of sleep apnea in shelter residents. | up to 4 years.
  Understanding the prevalence of sleep apnea in people experiencing homelessness
Changes of FOSQ-10 as an indicator of sleep-related quality of life score over the course of treatment period | 3 and 6 month after starting the treatment
  Understanding the effect of providing treatment on different aspects of quality of life
The effect of sleep apnea treatment on blood pressure in people experiencing homelessness | 3 and 6 month after starting the treatment
  Understanding the potential impact of sleep apnea treatment on blood pressure (as an index of cardiorespiratory condition)
Contributing factors to adherence rate (number of nights with treatment usage >4 hours / total number of nights monitored) at months 3 and 6 post-treatment. | 3 and 6 month after starting the treatment
  To investigate the factors that affect the adherence to preferred sleep apnea treatment in people experiencing homelessness

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Dixon Hall, Toronto, Ontario
  - Fred Victor, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
The data contains sensitive information about the participants and data sharing with the teams outside of the University Health Network has never been considered in consents obtained from participants.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT06620601/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT06620601/ICF_001.pdf